CLINICAL TRIAL: NCT02746679
Title: Impact of Mindfulness Based Stress Reduction on Anxiety, Depression and Quality of Life in Women With Intrauterine Adhesion:a Randomized Controlled Trial.
Brief Title: Impact of Mindfulness Based Stress Reduction on Anxiety, Depression and QOL in Women With Intrauterine Adhesion.
Acronym: IMBSRADQWIUA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuqing Chen (Other)
Responsible Party: Sponsor-Investigator, Yuqing Chen, associate professor, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MBSR-5
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Results first posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-05

CONDITIONS: Asherman Syndrome
Keywords: Asherman syndrome; Mindfulness; Anxiety; Depression; Quality of Life
MeSH Terms: conditions — Gynatresia; Anxiety Disorders; Depression | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBSR Group (Experimental): The Mindfulness Based Stress Reduction program consisted of eight weekly sessions, each 2.5 hours long, and delivered on consecutive weeks.The Mindfulness Based Stress Reduction therapist participated in the mindfulness exercises with group members during the weekly sessions, and group members were instructed to practice these mindfulness exercises outside group meetings for at least 45 minutes per day, 6 days per week.Group members were taught three main varieties of mindfulness skills: the body scan exercise, sitting meditation, and yoga exercises.The daily homework exercises consisted of repeating body scan work, sitting meditation and yoga exercises at home to provide practice and generalization of the skills.
  Interventions: Other: Mindfulness Based Stress Reduction
- wait-list control group (No Intervention): The patients assigned to the wait-list control group did not receive MBSR intervention for 8 weeks when participants in MBSR were engaged in the MBSR intervention.They only received conventional therapy.

INTERVENTIONS:
Other: Mindfulness Based Stress Reduction — Mindfulness Based Stress Reduction programs have been shown to be effective, however, the potential benefits of Mindfulness Based Stress Reduction to decrease depression, anxiety, stress in other diseases. Therefore, the purpose of this study was to examine whether MBSR is effective, and has potential as an intervention to decrease depression, anxiety ,and to improve quality of life of intrauterine adhesion patients.
  Arms: MBSR Group

SUMMARY:
The purpose of this study is to determine whether mindfulness based stress reduction are effective on improve anxiety, depression and quality of life in women with intrauterine adhesion

DETAILED DESCRIPTION:
This is a parallel arm, randomized controlled trials, according to 1: 1 ratio assigned intrauterine adhesions patients to mindfulness based stress reduction group and wait-list control group.The study compared anxiety and depression levels and quality of life in patients with intrauterine adhesions before and after the completion of mindfulness based stress reduction program.Anxiety, depression and quality of life level measured by the Zung self-rating anxiety scale, Zung Self-Rating Depression Scale and The 36-item Short-Form Health Survey.

ELIGIBILITY:
Inclusion Criteria:

1. Meet intrauterine adhesions diagnostic criteria of ESGE.
2. Patients with clear consciousness, can correct understanding related content of the questionnaire.

Exclusion Criteria:

1. Have a history of mental illness.
2. Receiving psychological treatment currently.
3. Have acute mental disorders.
4. Experienced special stress life events within six months.

Ages: 20 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 226 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuzhong Yao, professor, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Roth B, Robbins D. Mindfulness-based stress reduction and health-related quality of life: findings from a bilingual inner-city patient population. Psychosom Med. 2004 Jan-Feb;66(1):113-23. doi: 10.1097/01.psy.0000097337.00754.09. PMID 14747645
- [Background] Wurtzen H, Dalton SO, Elsass P, Sumbundu AD, Steding-Jensen M, Karlsen RV, Andersen KK, Flyger HL, Pedersen AE, Johansen C. Mindfulness significantly reduces self-reported levels of anxiety and depression: results of a randomised controlled trial among 336 Danish women treated for stage I-III breast cancer. Eur J Cancer. 2013 Apr;49(6):1365-73. doi: 10.1016/j.ejca.2012.10.030. Epub 2012 Dec 19. PMID 23265707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited into present study between January 2015 and January 2016
Pre-assignment Details: A total of 226 patients with IUA were recruited into present study within 12 months. Of them, 10 met the exclusion criteria and 55 patients refused to participate in this study. Finally, 161 patients were randomized into MBSR group (n=80) and wait-list group (n=81).
Groups:
- MBSR Group: The Mindfulness Based Stress Reduction program consisted of eight weekly sessions, each 2.5 hours long, and delivered on consecutive weeks.The Mindfulness Based Stress Reduction therapist participated in the mindfulness exercises with group members during the weekly sessions, and group members were instructed to practice these mindfulness exercises outside group meetings for at least 45 minutes per day, 6 days per week.Group members were taught three main varieties of mindfulness skills: the body scan exercise, sitting meditation, and yoga exercises.The daily homework exercises consisted of repeating body scan work, sitting meditation and yoga exercises at home to provide practice and generalization of the skills.
  Mindfulness Based Stress Reduction: Mindfulness Based Stress Reduction programs have been shown to be effective, however, the potential benefits of Mindfulness Based Stress Reduction to decrease depression, anxiety, stress in other diseases. Therefore, the purpose of this
Period: Overall Study
Arm/Group | MBSR Group | Wait-list Control Group
Started | 80 | 81
Completed | 76 | 75
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBSR Group | Wait-list Control Group | Total
Number analyzed (Participants) | 76 | 75 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (5.5) | 31.1 (6.5) | 30.9 (6.0)
Sex/Gender, Customized [Number; unit: participants]
  female | 76 | 75 | 151
Education [Number; unit: participants]
  ≥9 years | 71 | 67 | 138
  < 9 years | 5 | 8 | 13
Marriage [Number; unit: participants]
  Single | 12 | 7 | 19
  Married | 64 | 68 | 132
Salary per month [Number; unit: participants]
  < ¥ 5000 | 16 | 15 | 31
  > ¥ 5000 | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: The Zung Self-Rating Anxiety Scale Scores Before and After the Intervention
Description: The full name of the scale called Zung Self-Rating Anxiety Scale.The ZSAS contains 20 questions. Each question is scored on a scale of 1-4 (never, some of the time, relatively often, most of the time). Fifteen questions involve the assessment of increasing anxiety levels, and five questions involve decreasing anxiety levels.Each items points accumulated as raw scores,the lowest raw score is 20 points, the highest raw score is 80 points. The raw scores multiply by 1.25, taking the integer part as the standard scores.The ZSAS standard scores were used to define four categories of anxiety severity: within normal rangeor no significant psychopathology (25-49points);presence of mild to moderate anxiety levels (50-59points); severe anxiety levels (60-69points); and presence of extreme depression (70-100points).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(raw scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(raw scores)
  before intervention | 36.4 (6.2) | 37.3 (6.8)
  after intervention | 32.1 (5.9) | 38.5 (6.4)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p < 0.001, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

2. Secondary Outcome: Endometrial Thickness Were Measured by Ultrasound in the Middle of Menstruation in All Patients.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
mm
  before intervention | 4.4 (2.5) | 4.1 (2.4)
  after intervention | 5.7 (1.4) | 5.2 (1.4)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p > 0.05, ANOVA

3. Secondary Outcome: Menstruation Was Evaluated With Visual Analogue Scale (VAS) in Which the Menstruation Was Assessed by the Patients Themselves With 0 as Amenorrhea and 100 as Normal Menstruation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale
  before intervention | 43.9 (22.5) | 44.8 (27.8)
  after intervention | 68.5 (22.0) | 69.2 (24.8)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Numbers of Participants With Reformation of Intrauterine Adhesions Were Counted by the Follow-up Hysteroscopy Was Performed in the Third Month After the Surgery
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
participants
  Reformation of intrauterine adhesions | 14 | 26
  Normal uterine | 62 | 49
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.024, Chi-squared

5. Secondary Outcome: The Zung Self-Rating Depression Scale Scores Before and After the Intervention
Description: The full name of the scale called Zung Self-Rating Depression Scale.The ZSDS includes 10 positively worded items and 10 negatively worded items that assess symptoms of depression. Item responses are ranked from 1 to 4, and higher scores correspond to more frequent symptoms. For each item,patients give a score according to whether the item has occurred: 1 = never/very rarely; 2 = once in a while/some of the time/occasionally; 3 = relatively often/very often/often; 4 = most of the time/always. Each items points accumulated as raw scores,the lowest raw score is 20 points, the highest raw score is 80 points. The raw scores multiply by 1.25, taking the integer part as the standard scores.The ZSDS standard scores were used to define four categories of depression severity: within normal range or no significant psychopathology (below 51points); presence of minimal to mild depression (51-60points); presence of moderate to marked depression (61-70points).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(raw scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(raw scores)
  before intervention | 40.3 (7.2) | 39.7 (6.2)
  after intervention | 37.1 (7.4) | 40.9 (6.0)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p < 0.001, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

6. Secondary Outcome: The Scores of Physical Function Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: The 36-item Short-Form Health Survey (SF-36) is a commonly used generic questionnaire that includes 36 items clustered into eight dimensions (bodily pain, general health, mental health, physical functioning,role-emotional, role-physical, social functioning, and vitality). The item scores for each dimension are coded, summed and transformed to a scale from 0(worst possible health status) to 100 (best possible health status). Each raw scale score is linearly transformed to t scores. The transformed scores range from 0 to 100; higher scores indicate a better health-related QoL.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 86.5 (13.7) | 88.1 (12.5)
  after intervention | 90.9 (10.7) | 85.3 (11.3)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.001, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

7. Secondary Outcome: The Scores of Role-physical Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 61.5 (38.2) | 60.3 (35.9)
  after intervention | 74.7 (26.6) | 55.7 (34.3)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.003, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

8. Secondary Outcome: The Scores of Role-emotional Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 55.7 (34.3) | 64.0 (35.0)
  after intervention | 78.5 (22.9) | 62.7 (30.0)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.024, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

9. Secondary Outcome: The Scores of Vitality Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 67.2 (19.5) | 64.5 (19.8)
  after intervention | 74.9 (11.6) | 62.3 (18.6)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.004, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

10. Secondary Outcome: The Scores of Mental Health Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 64.6 (16.3) | 64.9 (16.8)
  after intervention | 72.9 (13.0) | 63.9 (16.5)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p < 0.001, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

11. Secondary Outcome: The Scores of Social Functioning Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 78.1 (19.6) | 80.3 (18.0)
  after intervention | 86.2 (13.9) | 80.5 (18.6)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p < 0.001, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

12. Secondary Outcome: The Scores of Bodily Pain Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 71.3 (15.1) | 70.4 (16.3)
  after intervention | 72.5 (11.1) | 68.5 (14.6)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.277, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

13. Secondary Outcome: The Scores of General Health Before and After the Intervention(One Dimensions of the 36-item Short-form Health Survey)
Description: as for outcome 6
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale(t scores)
Arm/Group | MBSR Group | Wait-list Control Group
Number analyzed (Participants) | 76 | 75
units on a scale(t scores)
  before intervention | 56.9 (17.7) | 58.9 (19.0)
  after intervention | 66.5 (16.0) | 57.1 (17.6)
Statistical Analysis 1: Comparison: MBSR Group vs Wait-list Control Group; Test type: Superiority or Other; p = 0.001, ANOVA; The comparison of the change from baseline to 8 weeks later between MBSR Group and wait-list control group

ADVERSE EVENTS:
Arm/Group | MBSR Group | Wait-list Control Group
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes